CLINICAL TRIAL: NCT05012488
Title: Comparison of the Effects of Morton's Neuroma on Foot Pressure Distribution and Gait Parameters in Pes Planus and Pes Cavus Patients
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Assistant Professor, Acibadem University
Other Study IDs: ATADEK 2021- 09/58
Record Dates: First submitted 2021-07-08; First posted 2021-08-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Morton Neuroma; Pes Planus; Pes Cavus
Keywords: gait; foot pressure
MeSH Terms: conditions — Morton Neuroma; Flatfoot; Talipes Cavus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morton Neuroma + pes planus: The effect of unilateral morton neuroma on gait parameters and foot pressure distribution in patients with bilateral pes planus will be investigated. Foot pressure distributions and gait parameters of the patients; foot rotation, step length, stance phase percentage, swing phase percentage, cadence, velocity, rerefoot pressure, midfoot pressure and forefoot pressure will be recorded with Zebris FDM -T ( Force distiribution Measurement Treadmill ) system. Zebris is a name of company in German .
  Interventions: Other: Comparison of gait and foot pressure
- Morton Neuroma + pes cavus: The effect of unilateral morton neuroma on gait parameters and foot pressure distribution in patients with bilateral pes cavus will be investigated. Foot pressure distributions and gait parameters of the patients; foot rotation, step length, stance phase percentage, swing phase percentage, cadence, velocity, rerefoot pressure, midfoot pressure and forefoot pressure will be recorded with Zebris FDM -T ( Force distiribution Measurement Treadmill ) system. Zebris is a name of company in German .
  Interventions: Other: Comparison of gait and foot pressure

INTERVENTIONS:
Other: Comparison of gait and foot pressure — The spatio temporal gait parameters of the patients will be evaluated with Zebris (Zebris Medical Limited , Germany) FDM (Force Distribution Measurement ) treadmill system. The system has production of 3D motion analysis and force measurement technologies for biomechanics. When the treadmill is in static and dynamic condition, strong pressure distribution measurement will be taken.

SUMMARY:
The aim of our study is to compare the effect of Morton's neuroma in feet with pes planus and pes cavus on foot pressure and temporal and spatial gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bilateral pes planus or pes cavus
* Diagnosis of unilateral Morton neuroma
* Confirmation of the diagnosis of Morton's neuroma with Magnetic Resonance Imaging (MRI)
* Pain level of the patients during walking is at least 3 according to the Visual Analogue Scale (VAS).

  * Volunteer to study over the age of 18

Exclusion Criteria:

* Having Symptomatic musculoskeletal disease in the lower extremity
* Having peripheral nervous system disease
* Presence of rigid deformity in the foot
* Extremity or contralateral extremity surgery with Morton's neuroma
* Having received physiotherapy in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients older than 18 years of age with bilateral pes planus or pes cavus accompanied by Morton's neuroma will be recruited by simple randomization.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Foot rotation | 4 weeks
  Foot rotation (degree), will be evaluated by Zebris (Zebris Medical Limited - Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system to assessment the angle between the longitudinal axis of the foot and the running direction. Negative value = inward rotation, positive value = outward rotation.Subtalar joint supination describes angulation in the negative direction and pronation describes the angulation in the positive direction.Unit of measure is degrees.
Step length | 4 weeks
  Step length (cm) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. Step length describes the distance between the heel contact of one side of the body and the heel contact of the contralateral side. Unit of measure is centimeter.
Stance phase percentage | 4 weeks
  Stance phase percentage (%) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Stance phase percentage describes the phase of a gait cycle in which the foot has contact with the ground.The unit is expressed as a percentage.
Swing phase percentage | 4 weeks
  Swing phase percentage (%) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Swing phase describes the phase of a gait cycle during which the foot has no contact with the ground. The unit is expressed as a percentage.
Cadance | 4weeks
  Cadence (steps/min) will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Cadence is steps/minute. It is defined as the step frequency.
Velocity | 4 weeks
  Velocity will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. The system measures average gait speed during the analyzed measuring interval. The unit is expressed as km/hr.
Foot pressure distiribution | 4 weeks
  Foot pressure distiribution will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. The system evaluate the average maximum values reached in N/cm² for the three zones: toes, mid-foot and heel.

SECONDARY OUTCOMES:
Demographic data/patient age | 4 weeks
  The ages of the patients will be recorded in the evaluation form.
Demographic data/patient weight | 4 weeks
  The weight of the patients will be recorded in the evaluation form in kilograms.
Demographic data/patient height | 4 weeks
  The height of the patients will be recorded in the evaluation form in meters.
Demographic data/patient body mass index BMI | 4 weeks
  The BMI of the patients will be recorded in the evaluation form in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Fulya Foot Surgery Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No